CLINICAL TRIAL: NCT00883870
Title: A Randomized, Double Blind, Multicentric, Placebo Controlled, Single Dose, Phase - i/ii Study Assessing the Safety and Efficacy of Intramuscular ex Vivo Cultured Adult Allogenic Mesenchymal Stem Cells in Patients With Critical Limb Ischemia (Cli)
Brief Title: Mesenchymal Stem Cells in Critical Limb Ischemia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Stempeutics Research Pvt Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SRPL/CLI/07-08/001
Record Dates: First submitted 2009-04-17; First posted 2009-04-20 (Estimated); Last update posted 2013-03-05 (Estimated); Status verified 2013-03

CONDITIONS: Critical Limb Ischemia
Keywords: mesenchymal stem cells; critical limb ischemia
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia | interventions — Plasmalyte A

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- mesenchymal stem cells (Experimental): Intramuscular injection
  Interventions: Drug: mesenchymal stem cells
- Placebo (Experimental): Intramuscular injection
  Interventions: Drug: Plasmalyte A

INTERVENTIONS:
Drug: mesenchymal stem cells — Intramuscular injection
  Arms: mesenchymal stem cells
Drug: Plasmalyte A — Intramuscular injection
  Arms: Placebo

SUMMARY:
This clinical trial aims to study the safety and efficacy of adult mesenchymal stem cells in critical limb ischemia.

ELIGIBILITY:
Inclusion Criteria:

* Males or females with non-child bearing potential in the age group of 18-60 yrs of Indian origin.
* Established CLI, clinically and hemodynamically confirmed as per Rutherford- II-4, III-5, or III-6; Patients having Infra-inguinal arterial occlusive disease with rest pain or ischemic ulcer/necrosis, who are not eligible for or have failed traditional revascularization treatment (No option patients)
* Ankle Brachial Pressure Index (ABPI) ≤ 0.6 or ankle pressure ≤ 70 mm Hg or TcPO2 ≤ 60 mmHg in the foot
* Patients if having associated Type II Diabetes, should be on medication and well controlled (HbA1c ≤ 8%) without complications
* Patients who are able to understand the requirements of the study, and willing to provide voluntary written informed consent, abide by the study requirements, and agree to return for required follow-up visits
* Normal liver and renal function
* On regular medication for hypertension if any

Exclusion Criteria:

* Patients with CLI suitable for surgical or percutaneous revascularization as determined by the surgeon performing vascular procedure and patients with any acute/chronic inflammatory condition
* CLI patient requiring amputation proximal to trans-metatarsal level
* Patients with gait disturbance for reasons other than CLI.
* Type I diabetes
* Patients having respiratory complications/left ventricular ejection fraction < 25%f) Stroke or myocardial infarction within last 3 months
* Patients who are contraindicated for MRA
* Have clinically serious and/or unstable inter-current infection, medical illnesses or conditions that are uncontrolled or whose control, in the opinion of the Investigator, may be jeopardized by participation in this study or by the complications of this therapy
* Documented terminal illness or cancer or any concomitant disease process with a life expectancy of less than 1 year
* Patients already enrolled in another investigational drug trial or completed within 3 months.
* History of severe alcohol or drug abuse within 3 months of screening.
* Hb% < 10 gm%, Serum Creatinine ≥ 2mg%, Serum Total Bilirubin ≥2mg%, HbA1c > 8%
* Women with child bearing potential, pregnant and lactating women.
* Patients tested positive for HIV 1, HCV, HBV,

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2009-04; Primary Completion 2010-02 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
AE and symptomatic relief | 6 months

SECONDARY OUTCOMES:
Increase in transcutaneous partial oxygen pressure (TcPO2) and Ankle brachial pressure index (ABPI) - measured by Doppler | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Suresh K R, Principal Investigator — Bhagawan Mahaveer Jain Heart Centre, Bangalore; Sanjay Desai, Principal Investigator — M.S.Ramaiah Memorial Hospital, Bangalore; Rajiv Parakh, Principal Investigator — Sri Ganga Ram Hospital, New Delhi; Sudhindran S, Principal Investigator — Amrita Institute of Medical Sciences, Kochi
Locations (4):
- India (4):
  - M.S.Ramaiah Memorial Hospital, Bangalore, Karnataka
  - Bhagawan Mahaveer Jain Heart Centre, Bangalore, Karnataka
  - Amrita Institute of Medical Sciences, Kochi, Kerala
  - Sri Ganga Ram Hospital, New Delhi, New Delhi

REFERENCES:
- [Derived] Gupta PK, Chullikana A, Parakh R, Desai S, Das A, Gottipamula S, Krishnamurthy S, Anthony N, Pherwani A, Majumdar AS. A double blind randomized placebo controlled phase I/II study assessing the safety and efficacy of allogeneic bone marrow derived mesenchymal stem cell in critical limb ischemia. J Transl Med. 2013 Jun 10;11:143. doi: 10.1186/1479-5876-11-143. PMID 23758736